CLINICAL TRIAL: NCT06225583
Title: Precise and Objective Identification of Bertolotti Syndrome Using Novel Kinematic Biomarkers
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Steinmetz, MD, Chairman, Department of Neurosurgery, The Cleveland Clinic
Other Study IDs: IRB 22-1310
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Bertolotti's Syndrome; Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bertolotti's Syndrome: Subjects with Bertolotti's Syndrome.
- Non-Bertolotti's Lower Back Pain: Subjects without Bertolotti's Syndrome with lower back pain.

SUMMARY:
The purpose of this study is to collect lumbar rotations, velocity, and accelerations, along with pain scores using a novel dynamic VAS device, from twenty (20) Bertolotti Syndrome patients and twenty (20) non-Bertolotti low back pain patients during range-of-motion tasks. The assessments will be analyzed to determine the differences in kinematics and continuous pain scores between Bertolotti patients and non-Bertolotti low back pain patients.

ELIGIBILITY:
Inclusion Criteria:

Lower Back Pain Cohort

* Positive diagnosis of sacroiliac pain or lumbosacral facet arthritis pain
* Age ≥ 18 years

Bertolotti's Syndrome Cohort

* Positive diagnosis of Bertolotti's Syndrome
* Age ≥ 18 years
* Positive imaging for Bertolotti's Syndrome
* Previous analgesic injection results

Exclusion Criteria:

Lower Back Pain Cohort

* History of spinal deformity, previous spinal surgeries, spinal infections
* Pregnant women

Bertolotti's Syndrome Cohort

* History of spinal deformity, previous spinal surgeries, spinal infections
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 Bertolotti's Syndrome patients and 20 lower back pain patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify Bertolotti's Syndrome-specific kinematic biomarkers using collected patient kinematic and real-time VAS data from range-of-motion tasks. | 2025

CONTACTS AND LOCATIONS:
Overall Officials: Michael Steinmetz, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States